CLINICAL TRIAL: NCT00470860
Title: Educational Technology to Enhance Diabetes Care - Retention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: G04-07-038-02
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Participation in LOFTS online tutorial

SUMMARY:
This study mapped the time course of forgetting among resident physicians after they use an online learning exercise covering principles of diabetes care. Participants took a pre-test followed by an online tutorial covering aspects of diabetes care. They then completed a post-test on the same topics after a randomly-assigned time delay from 0 to 55 days. We hypothesized that post-test scores after these different time delays would decline following a curvilinear relationship with increasing time. This understanding of forgetting will inform our selection of a time for delivering reinforcement exercises in future educational studies among physicians.

ELIGIBILITY:
Inclusion Criteria:

* Family medicine residents (physicians in training)
* Internal medicine residents (physicians in training)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2004-12; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Knowledge related to blood pressure and lipid management for diabetes patients | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Bell, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Charles R. Drew University, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California